CLINICAL TRIAL: NCT06555705
Title: Effect of Omega 3 Supplementation on the Heart Rate Variability in Obese Children, a Clinical Trial
Brief Title: Effect of Omega 3 Supplementation on the Heart Rate Variability in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Atef Abdelsattar Ibrahim, Lectuere of Pediatrics and Pediatric Clinical Nutrition, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-547-2023
Record Dates: First submitted 2024-08-11; First posted 2024-08-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group recieveing omega 3 and the standard nutritional regimen for 3 months (Experimental): The intervention group will be examined by 10 -minutes Holter and then omega 3 will be given to children( at least 400 mg eicosapentaenoic acid (EPA) and 120 mg docosahexaenoic acid (DHA) daily in addition to the standard nutritional regimen ) daily for 3 months and then reassesent of Holter will be carried out .
  Interventions: Dietary Supplement: Omega 3
- Control group receiving placebo and the standard nutritional regimen for 3 months (Placebo Comparator): The control group will be examined by 10 -minutes Holter and then the standard nutritional regimen will be given daily for 3 months and then reassessment of Holter will be carried out .
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — The control group will be given placebo for 3 months
  Arms: Control group receiving placebo and the standard nutritional regimen for 3 months
Dietary Supplement: Omega 3 — The interventional group will be given omega 3 for 3 months
  Arms: Interventional group recieveing omega 3 and the standard nutritional regimen for 3 months

SUMMARY:
Evidence shows that omega-3 fatty acids lower blood triglyceride levels, lower blood pressure, enhance insulin sensitivity, and improve heart rate variability (HRV) measures, all of which may be indicators of cardiovascular health.As a result, omega-3 fatty acid supplementation may be a low-cost strategy with little adverse effects for obese youngsters, perhaps delaying the development of chronic cardiovascular illnesses.

DETAILED DESCRIPTION:
This is a two-armed study , the interventional group will be given omega 3 and the control group will be given a placebo and both will be examined for the heart rate variability

ELIGIBILITY:
Inclusion Criteria:

* Children (5-12 years) whose parents or caregivers will agree to be enrolled in the study
* Obese Children (Simple obesity )
* Both males and females

Exclusion Criteria:

* Patients are known to have cardiac disease
* Patients with associated chronic systemic illness
* Patients with 2ry obesity : (endocrine /metabolic/genetics/drug intake)
* Patients on medications affecting heart rate :structural or arrhythmic

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
The effect of omega-3 on heart rate variability that is represented in the root mean square of successive differences of the heart rates ( RMSSD ) in obese children | 3 months
  Obese children will be examined for the effect of Omega-3 supplementation on heat rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Rodina Sobhy, Study Director — Professor of Pediatrics
Locations (1):
- Hoda Atef Abdelsattar Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Throughout the study, the privacy and confidentiality of the data will be perceived, the results will be presented anonymously without disclosure of patients' personal identifying information.